CLINICAL TRIAL: NCT00500539
Title: An Open Label, Single Arm Study to Assess the Safety and Immunogenicity of Omalizumab Liquid Administered Subcutaneously to Male and Female Adolescents and Adults With Persistent Allergic Asthma
Brief Title: Open Label Study to Assess Safety and Immunogenicity of Omalizumab Liquid Formulation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Genentech, Inc. (Industry); Tanox (Industry)
Responsible Party: external affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025C2303
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
Keywords: Asthma; omalizumab; safety; allergic asthma; adolescents
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: omalizumab — The liquid formulation of omalizumab was packaged in a pre-filled safety syringe containing either 75 mg (0.5ml) or 150 mg (1.0 ml) of drug. The syringes were clearly marked so that the health care provider could differentiate between the 75 mg or 150 mg syringe.

SUMMARY:
The primary objective of this study is to assess the immunogenic potential of the liquid formulation of omalizumab administered over a period of 6 months in moderate to severe persistent allergic asthma patients 12 years of age or older, with no previous exposure to the drug (omalizumab naïve patients). The secondary objective of this study is to assess the safety of the liquid formulation of omalizumab in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 12 years old or above with moderate to severe allergic asthma
* Body weight greater than 30kg and less than 150 kg and total serum IgE level greater than 30 to less than 700 IU/ml
* Diagnosis of allergic asthma greater than 1 year duration, according to the American Thoracic Society criteria (14) and at screening, a history consistent with clinical features of moderate to severe persistent asthma.
* Positive skin prick test (diameter of wheel is greater than 3mm) to at least one perennial allergen within the previous one year to visit 1, to which the patient will be exposed on a regular basis (most days) for the duration of the study.
* No clinically significant asthma exacerbations that required treatment with systemic corticosteroids during the four weeks immediately prior to screening visit (Visit 1) and during screening period (between Visit 1 and 2)
* Demonstrated evidence of inadequate asthma symptom control, despite treatment with ICS according to clinical features of moderate to severe persistent asthma.

Exclusion Criteria:

* Previous exposure to omalizumab
* Previous exposure to other humanized proteins or monoclonal antibodies
* Known HAHA to other monoclonal antibodies
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* Known hypersensitivity to any ingredients, including excipients of the study medication or drugs related to omalizumab (e.g. monoclonal antibodies, polyclonal gamma globulin)
* Active lung disease other than allergic asthma (e.g. cystic fibrosis, bronchiectasis)
* Elevated serum IgE levels for reasons other than allergy (e.g. parasite infections, hyperimmunoglobulin E syndrome, Wiskott-Aldrich Syndrome or allergic bronchopulmonary aspergillosis)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bardelas, MD, Principal Investigator — Allergy and Asthma center of North Carolina, PA, High Point, NC 27262
Locations (31):
- United States (26):
  - Allergy & Immunology Associates, Ltd, Scottsdale, Arizona
  - California Allergy and Asthma Medical Group, Palmdale, California
  - Allergy Associates Medical Group, Inc,, San Diego, California
  - Bensch Research Associates, Stockton, California
  - 1st Allergy and Clinical Research Center, Centennial, Colorado
  - Innovative Research of West Florida, Inc., Largo, Florida
  - Georgia Pollen, Albany, Georgia
  - Kansas City Allergy & Asthma, Overland Park, Kansas
  - Asthma and Allergy Specialists, PA, Minneapolis, Minnesota
  - : The Clinical Research Center, LLC, St Louis, Missouri
  - Allergy, Asthma and Clinical Immunology, Brick, New Jersey
  - Asthma & Allergy Research of NJ, Inc., Mount Laurel, New Jersey
  - Nassau Chest Pysicians, PC, Massapequa, New York
  - Allergy and Asthma Center of NC, PA, High Point, North Carolina
  - Allergy Center at Brookstone, Columbus, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Asthma and Allergy Center, Toledo, Ohio
  - The Corvallis Clinic, PC, Corvallis, Oregon
  - Allergy, Asthma & Dermatology Research Center, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy & Asthma Specialists, PC, Blue Bell, Pennsylvania
  - Asthma Allergy & Pulmonary Associates, PC, Philadelphia, Pennsylvania
  - AAPRI Clinical Research Institute, Providence, Rhode Island
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Allergy and Asthma Associates, Houston, Texas
  - Clinical Trials of North Houston, Houston, Texas
- Argentina (4):
  - Novartis Investigative Site,, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site,, Corrientes
  - Novartis Investigative Site,, Mendoza
- Novartis Investigator site, Nuremberg, Germany

REFERENCES:
- [Derived] Somerville L, Bardelas J, Viegas A, D'Andrea P, Blogg M, Peachey G. Immunogenicity and safety of omalizumab in pre-filled syringes in patients with allergic (IgE-mediated) asthma. Curr Med Res Opin. 2014 Jan;30(1):59-66. doi: 10.1185/03007995.2013.844115. Epub 2013 Oct 1. PMID 24028677

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab: The determined dose was injected subcutaneously every 2 weeks or every 4 weeks. Dose and dosing interval were determined based on patient body weight and pre-treatment serum IgE level; a dosing table was used.
Period: Treatment Period (24 Weeks)
Arm/Group | Omalizumab
Started | 155
Completed | 140
Not Completed | 15
Not completed — Adverse Event | 4
Not completed — Unsatisfactory therapeutic effect | 1
Not completed — Subject withdrew consent | 1
Not completed — Lost to Follow-up | 2
Not completed — Administrative problems | 2
Not completed — Protocol Deviation | 5
Period: Follow-up Period (16 Weeks)
Arm/Group | Omalizumab
Started | 148 (Participants could discontinue study drug and still enter the follow-up period.)
Completed | 136
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Subject withdrew consent | 2
Not completed — Lost to Follow-up | 3
Not completed — Administrative problems | 1
Not completed — Death | 1
Not completed — Protocol Deviation | 1
Not completed — Missing | 3

BASELINE CHARACTERISTICS:
Arm/Group | Omalizumab
Number analyzed (Participants) | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 135
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 42.7 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Confirmed Positive Human Antihuman Antibody (HAHA) Results at the End of the 16-week Follow-up Period
Description: An assessment of the immunogenic potential of omalizumab liquid was a primary objective of the study, and was based on the results of the human anti-human antibody (HAHA) assays at the end of the follow-up period. A participant was considered potentially HAHA positive if either Fab or Fc was more than 2.0 titer. All values more than 2.0 titer were re-assayed to obtain a confirmatory result. Confirmatory results were used to determine those participants who were HAHA positive.
Time Frame: 16 weeks after last dose
Population: The Safety Population consisted of all patients that received any part of a dose of study drug and had any post-baseline assessment, whether scheduled or not. The analysis was done on total number of patients who had follow-up HAHA sample taken.
Measure: Number; unit: participants
Groups:
- Follow-up Period: Participants were evaluated at 16 weeks after the last dose of study drug.
Arm/Group | Follow-up Period
Number analyzed (Participants) | 136
participants
  Fab HAHA Positive - Negative at baseline | 0
  Fab HAHA Positive - Positive at baseline | 0
  Fab HAHA Positive - Missing at baseline | 0
  Fc HAHA Positive - Negative at baseline | 0
  Fc HAHA Positive - Positive at baseline | 0
  Fc HAHA Positive - Missing at baseline | 0
  Fab and/or Fc HAHA Positive - Fab and Fc HAHA -Ve | 0
  Missing at baseline | 0

2. Secondary Outcome: Number of Participants Who Experienced Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Treatment Period
Description: The assessment of safety was based on the number of patients with AEs (mild, moderate and severe) and SAEs. According to FDA 21CFR 314.80, a serious adverse event (SAE) is described as any adverse event that leads to death, is life threatening, causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event not described above. The duration of the treatment period was 24 weeks, but patients were followed for an additional 4 weeks, so that the total duration of the treatment period for purposes of AE reporting was 28 weeks.
Time Frame: 24 weeks treatment period + 4 weeks for following up participants
Population: The safety population consisted of all patients that received any part of a dose of study drug and had any post-baseline assessment, whether scheduled or not.
Measure: Number; unit: participants
Groups:
- Treatment Period: The determined dose was injected subcutaneously every 2 weeks or every 4 weeks. Dose and dosing interval were determined based on patient body weight and pre-treatment serum IgE level; a dosing table was used.
Arm/Group | Treatment Period
Number analyzed (Participants) | 155
participants
  Participants with AEs during the treatment period | 124
  Mild AEs | 25
  Moderate AEs | 76
  Severe AEs | 23
  AEs suspected to be related to study drug | 22
  AEs not suspected to be related to study drug | 102
  Deaths | 1
  Serious Adverse Events (SAEs) | 14
  Discontinued due to Adverse Events | 4
  Discontinued due to Serious Adverse Events | 2
  Discontinued due to non-serious Adverse Events | 2

3. Secondary Outcome: Number of Participants Who Experienced Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Follow-up Period
Description: The assessment of safety was based on the number of patients with AEs (mild, moderate and severe) and SAEs. According to FDA 21CFR 314.80, a serious adverse event (SAE) is described as any adverse event that leads to death, is life threatening, causes or prolongs hospitalization, results in a congenital anomaly, or any other important medical event not described above. The duration of the follow-up period was 16 weeks, but for purposes of AE reporting the follow-up period was 12 weeks (as the first 4 weeks of follow-up were included in the treatment period).
Time Frame: Last 12 weeks of the follow-up period (initial 4 weeks of the follow-up period were included in the treatment period for AE reporting)
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Follow-up Period: Participants were assessed at 16 weeks after the last dose of study drug
Arm/Group | Follow-up Period
Number analyzed (Participants) | 148
participants
  Participants with AEs during the follow-up period | 51
  Mild AEs | 11
  Moderate AEs | 37
  Severe AEs | 3
  AEs suspected to be related to study drug | 0
  AEs not suspected to be related to study drug | 51
  Deaths | 0
  Serious adverse events (SAEs) | 1
  Discontinued due to Adverse Events | 1
  Discontinued due to Serious Adverse Events | 0
  Discontinued due to non-serious Adverse Events | 1

ADVERSE EVENTS:
Time Frame: Treatment period AEs were collected from first treatment dose until 28 days post last treatment dose (28 weeks total). Follow-up period AEs defined as AEs that began after 28 days post last treatment dose until the end of the follow-up (12 weeks total).
Description: The safety population consisted of all patients that received any part of a dose of study drug and had any post-baseline assessment, whether scheduled or not.
Groups:
- Omalizumab Treatment Period: The determined dose was injected subcutaneously every 2 weeks or every 4 weeks. Dose and dosing interval were determined based on patient body weight and pre-treatment serum IgE level; a dosing table was used.
- Omalizumab Follow up Period: Participants were assessed at 16 weeks after the last dose of study drug
Arm/Group | Omalizumab Treatment Period | Omalizumab Follow up Period
Serious Adverse Events (participants affected / at risk) | 14/155 | 1/148
Other Adverse Events (participants affected / at risk) | 74/155 | 34/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab Treatment Period (N=155) | Omalizumab Follow up Period (N=148)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab Treatment Period (N=155) | Omalizumab Follow up Period (N=148)
Gastroenteritis viral (Infections and infestations) | 8 | 0
Nasopharyngitis (Infections and infestations) | 15 | 3
Sinusitis (Infections and infestations) | 27 | 12
Upper respiratory tract infection (Infections and infestations) | 18 | 6
Headache (Nervous system disorders) | 13 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 24 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or the publication of the trial results in their entirety.